CLINICAL TRIAL: NCT06983418
Title: Euthyroid Sick Syndrome in Severe Obesity Hypoventilation Patients Admitted to Intensive Care Unit; Incidence, Risk Factors and Outcome
Brief Title: Euthyroid Sick Syndrome in Obesity Hypoventilation Syndrome
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: R.21.08.1406
Record Dates: First submitted 2025-05-02; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2021-09

CONDITIONS: Euthyroid Sick Syndrome; Obesity Hypoventilation Syndrome (OHS)
Keywords: Euthyroid Sick Syndrome; Obesity Hypoventilation Syndrome; Acute Respiratory Failure
MeSH Terms: conditions — Euthyroid Sick Syndromes; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESS Group - OHS Patients with Euthyroid Sick Syndrome: Participants with Obesity Hypoventilation Syndrome (OHS) admitted to the intensive care unit (ICU) for acute hypercapnic respiratory failure who were diagnosed with Euthyroid Sick Syndrome (ESS). ESS was defined by low total triiodothyronine (TT3) levels, with or without low total thyroxine (TT4) and/or thyroid-stimulating hormone (TSH), measured within 24 hours of ICU admission.
- Non-ESS Group - OHS Patients without Euthyroid Sick Syndrome: Participants with Obesity Hypoventilation Syndrome (OHS) admitted to the ICU for acute hypercapnic respiratory failure who had normal thyroid function tests (TT3, TT4, and TSH) and did not meet criteria for Euthyroid Sick Syndrome, based on testing within 24 hours of ICU admission.

SUMMARY:
The goal of this observational study is to learn about the frequency and clinical impact of Euthyroid Sick Syndrome (ESS) in patients with Obesity Hypoventilation Syndrome (OHS) who are admitted to the intensive care unit (ICU) for acute respiratory failure.

The main question it aims to answer is:

How common is ESS in critically ill OHS patients, and does it affect the severity of illness and ICU outcomes?

Participants with OHS who are admitted to the ICU will have blood tests for thyroid hormone levels (TT3, TT4, and TSH) within 24 hours of admission. Researchers will compare illness severity, oxygen levels, need for breathing support, ICU stay duration, and outcomes between those with and without ESS.

DETAILED DESCRIPTION:
Obesity Hypoventilation Syndrome (OHS) is a serious respiratory condition that often requires ICU admission during acute decompensation. Emerging evidence suggests a potential link between systemic hypoxia and alterations in thyroid hormone levels, known as Euthyroid Sick Syndrome (ESS). While ESS is well documented in critical illness, its prevalence and clinical implications in the context of OHS remain poorly defined.

This prospective cross-sectional study was conducted in a tertiary ICU and enrolled adult patients admitted with acute respiratory failure attributed to OHS. The objective was to assess the prevalence of ESS and explore its association with clinical severity and ICU outcomes. Thyroid function tests, including total triiodothyronine (TT3), total thyroxine (TT4), and thyroid-stimulating hormone (TSH), were measured within 24 hours of ICU admission. ESS was defined by a low TT3 level, with or without reductions in TT4 and TSH, in the absence of known thyroid disease.

Additional data collected included arterial blood gas parameters, ventilatory support requirements (including non-invasive ventilation settings), and APACHE II scores. The study compared ICU course and outcomes, such as length of stay, need for invasive ventilation, and in-hospital mortality, between patients with and without ESS.

This study intends to clarify the clinical significance of thyroid dysfunction in OHS and examine whether ESS reflects a state of increased disease burden in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of Obesity Hypoventilation Syndrome (OHS), either pre-existing or newly established during ICU admission
* Admitted to the intensive care unit (ICU) with acute hypercapnic respiratory failure, defined as:

  * Arterial pH < 7.35
  * PaCO₂ > 45 mmHg
* Thyroid function tests performed within 24 hours of ICU admission
* Written informed consent provided by patient

Exclusion Criteria:

* Known history of thyroid disease (e.g., hypothyroidism, hyperthyroidism, thyroiditis, central hypothyroidism)
* Presence of acute conditions known to affect thyroid function tests, including:

  * Sepsis
  * Pneumonia
  * Active malignancy
  * Liver cirrhosis
  * Kidney failure
  * Heart failure
* Use of medications affecting thyroid function, including:

  * Corticosteroids
  * Amiodarone
  * Iodinated contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included adult patients (aged 18 years and older) with Obesity Hypoventilation Syndrome (OHS) who were admitted to the Intensive Care Unit (ICU) at Mansoura University Hospital in Mansoura, Egypt, for acute hypercapnic respiratory failure. Patients were enrolled between September 2021 and October 2023 and underwent thyroid function testing within 24 hours of ICU admission. The population was drawn from a tertiary care academic center serving a broad urban and rural population in the Nile Delta region.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
ICU Mortality | During ICU stay (assessed up to 28 days)

SECONDARY OUTCOMES:
ICU Length of Stay | Duration of ICU admission (assessed up to 28 days)
Need for Invasive Mechanical Ventilation | During ICU stay (assessed up to 28 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Mansoura University, Al Mansurah, Dakahlia/Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No